CLINICAL TRIAL: NCT00425139
Title: Multi-site Evaluation of a Video Game for Adolescents and Young Adults With Cancer
Brief Title: Evaluation of a Video Game for Adolescents and Young Adults With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HopeLab Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HL-04-001
Record Dates: First submitted 2007-01-19; First posted 2007-01-22 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2007-01

CONDITIONS: Neoplasms
Keywords: Cancer; Video game; Adolescent; Young adult
MeSH Terms: conditions — Neoplasms

INTERVENTIONS:
Behavioral: Re-Mission

SUMMARY:
The purpose of this study is to determine the effects of playing the interactive video game, Re-Mission, on patient outcomes, including adherence to medical treatment regimes, self-care behaviors, quality of life, stress, communication, control, and knowledge.

DETAILED DESCRIPTION:
POPULATION: Approximately 340 patients will be enrolled in this study. Patients will be 13 to 29 years of age with any cancer (original diagnosis or relapse), currently receiving treatment and expected to be on treatment for at least 4 - 6 months following Baseline assessment, and able to communicate effectively in English, Spanish, or French. Approximately 170 patients will be enrolled in each of the two treatment groups. Each group will receive either the "Re-Mission" video game and a popular interactive video game, or just the popular interactive video game.

DESIGN: This is a multi-center, randomized trial, with patients randomized to one of two groups. One group (50% of patients) will receive the active intervention, which is the psycho-educational video game module called Re-Mission and a popular video game (hereafter "RE-MISSION") and another group (50 % of patients) will be in a game control group and receive a popular video game only (hereafter "GAME CONTROL. The games in the RE-MISSION and GAME CONTROL groups are delivered on identical mini, personal computers (hereafter "Mini-PC").

INTERVENTION: Each patient in the RE-MISSION group will be asked to play "Re-Mission" along with the popular video game for at least one hour a week for a period of ten to fourteen weeks. "Re-Mission" presents a 3-D environment in which the player can manipulate a humanoid character inside the virtual body of a patient with cancer. Game-play consists of guiding the character to destroy cancer cells and other "enemies" in the body (e.g., bacteria) while avoiding injury or weakness. During the process of playing the game and guiding the character through a series of missions, the player learns about chemotherapy and other medical treatments, health-promoting self-care behaviors, infections, and pain management. In addition, the game has also been designed to facilitate the patient's ability to share knowledge and concerns with others.

DURATION OF STUDY: 9 -12 months

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient 13 to 29 years of age with a cancer diagnosis.
2. Patient who is currently receiving treatment and is expected to remain on treatment for at least 4 - 6 months.

Exclusion Criteria:

1. Patient who has a history of seizures due to photosensitivity.
2. Patient who has been determined by the investigator to be incapable of following the study schedule or study directions for any reason.
3. Patient who can not communicate effectively with study personnel in English, Spanish, or French.

Ages: 13 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 375
Dates: Start 2004-10; Study Completion 2005-11

PRIMARY OUTCOMES:
Adherence
Self-efficacy
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Pamela M Kato, Principal Investigator — HopeLab Foundation
Locations (34):
- United States (27):
  - City of Hope National Medical Center, Duarte, California
  - Los Angeles Children's Center for Cancer and Blood Disease, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital at Stanford, Palo Alto, California
  - Children's Hospital of SW Florida / Lee Memorial Health System, Fort Myers, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Children's Hospital of Tampa, Tampa, Florida
  - Kapiolani Medical Center, Honolulu, Hawaii
  - LSU Children's Hospital of New Orleans, New Orleans, Louisiana
  - Dana-Farber Cancer Institute and Children's Hospital, Boston, Massachusetts
  - DeVos Children's Hospital, Grand Rapids, Michigan
  - St John Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Children's Health Care - Minneapolis, Saint Paul, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - Washington University, St Louis, Missouri
  - Children's Hospital of New Mexico, Albuquerque, New Mexico
  - Golisano Children's Hospital, University of Rochester, Rochester, New York
  - Warren Clinic / Saint Francis Hospital, Tulsa, Oklahoma
  - Legacy Emanuel Children's Cancer Program, Portland, Oregon
  - Doernbecher Childrens Hospital - OHSU, Portland, Oregon
  - Children's Hospital of Austin, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Christus Santa Rosa Children's Hospital, San Antonio, Texas
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - Deaconess Medical Center, Spokane, Washington
- Royal Children's Hospital, Parkville, Victoria, Australia
- Canada (6):
  - Calgary Alberta Children's Hospital, Calgary, Alberta
  - McMaster University, Hamilton, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - McGill Univ Health Ctr - Montreal Children's Hospital, Montreal, Quebec
  - Hôpital Ste-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Québec, Ste-Foy, Quebec

REFERENCES:
- [Derived] Kato PM, Cole SW, Bradlyn AS, Pollock BH. A video game improves behavioral outcomes in adolescents and young adults with cancer: a randomized trial. Pediatrics. 2008 Aug;122(2):e305-17. doi: 10.1542/peds.2007-3134. PMID 18676516
- See also: Sponsor's website — http://www.hopelab.org
- See also: video game website — http://www.re-mission.net